CLINICAL TRIAL: NCT07023445
Title: Patterns of Inclisiran Use in the Real World: A Retrospective Analysis of US Databases
Brief Title: Patterns of Inclisiran Use in the Real World: An Analysis of US Databases
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839D1US01
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Atherosclerotic Cardiovascular Disease; Familial Hypercholesterolemia
Keywords: Low-density lipoprotein cholesterol; Real-world
MeSH Terms: conditions — Atherosclerosis; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Inclisiran Cohort: Patients with a prescription or claim for inclisiran.
- Alirocumab Cohort: Patients with a prescription or claim for alirocumab.
- Evolocumab Cohort: Patients with a prescription or claim for evolocumab.

SUMMARY:
This was a retrospective observational cohort study of patients who initiated inclisiran, alirocumab, or evolocumab in a real-world setting in the United States. The study used data extracted from three databases: (1) open and closed claims from Komodo's Healthcare map and electronic medical records (EMRs) from outpatient clinics affiliated with (2) Healix and (3) Metro Infusion Centers.

The study period spanned from 01 January 2021 to the latest date of the available data for each database. Index date was defined as the date of the first claim for inclisiran, alirocumab, or evolocumab within the patient identification period. The 12-month period prior to the index date (including the index date) was the baseline period. Follow-up spanned from the index date up to patient disenrollment, death, or the end of the study period, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first claim for inclisiran within the identification period.
* Patients without a claim for inclisiran and with a first alirocumab claim or first evolocumab claim within the identification period.
* Patients with 12 months of continuous enrollment (CE) before index, inclusive of index date.

Additional inclusion criteria for secondary outcome measures:

* Patients with at least 6-month or 12-month CE period post-index.
* Patients with continuous use of the index medications.
* Patients with available low-density lipoprotein cholesterol (LDL-C) measurements at baseline and after treatment initiation.

Exclusion criteria:

• Patients with ≥1 prescription claims for the index medications in the 12-month prior-index period (exclusive of index date).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 37688 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients per Demographic Category | Baseline
  Demographics included:
  * Age group
  * Gender
  * Insurance type
  * Race/ethnicity
Number of Patients per Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * Body mass index
  * Atherosclerotic Cardiovascular Disease (ASCVD) diagnosis
  * Familial Hypercholesterolemia (FH) diagnosis
  * Comorbidities
  * Type of lipid lowering therapy (LLT)

SECONDARY OUTCOMES:
Change From Baseline in LDL-C Levels | From Baseline up to 1 year
Number of Patients who Achieved a Reduction of 50% or more in LDL-C Levels After Initiating Treatment | Up to 1 year
Number of Patients who Achieved LDL-C Levels Below 70 Milligrams per Deciliter (mg/dL) and 55 mg/dL After Initiating Treatment | Up to 1 year
Medication Adherence | Up to 1 year
  Adherence was defined using proportion of days covered (PDC) within a period that the patient was persistent: the number of days covered by the prescription fills divided by the number of days between the first fill of the medication during the identification period (index date) and the end of the observational period. A patient was classified as having poor adherence if the calculated PDC was below 80%.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States